CLINICAL TRIAL: NCT02519894
Title: Effect of Intensive Low Sodium Restriction on Glomerular Infiltration Rate in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: PANTHITA SORNHIRAN (Other)
Responsible Party: Sponsor-Investigator, PANTHITA SORNHIRAN, PANTHITA SORNHIRAN, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Ramathibodi Hospital
Record Dates: First submitted 2015-08-09; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Declination of Glomerular Infiltration Rate in Chronic Kidney Disease Population

ARMS (2):
- Intervention group (Experimental): Intensive low sodium education and immediate sodium intake feedback by dietary scanning calculator
  Interventions: Behavioral: Dietary Scanning Calculator
- Controlled group (Placebo Comparator): Standard education

INTERVENTIONS:
Behavioral: Dietary Scanning Calculator
  Arms: Intervention group

SUMMARY:
Introduction :

Due to Chronic kidney disease is a public health problem, which is important increased in both developed and developing countries . And sodium intake restriction was related to the reduction of blood pressure and urine protein which is one of the important risk factor in chronic kidney disease. One of the problem in sodium restriction failure in Thai population with CKD nowadays is lack of knowledge and problem unawareness.

The study hypothesis :

Intense knowledge about sodium reduction and immediate feedback of the sodium intake could be simultaneously modifying the behavior to reduce sodium intake , blood pressure and also GFR reduction rate

Objectives :

To compare the effect of dietary salt restriction on glomerular filtration rate (GFR) between CKD patients receiving strict controlled combined with immediate individual feedback (DISC Progrram) and those receiving standard education.

Study design :

Multicenter, open labeled, parallel, randomized controlled trial

Sample size : 600

Primary outcome : GFR reduction (CKD-EPI)

Secondary outcome :

* Achievement rate of Na intake < 2 g/day (Urine Na < 90 mEq/day)
* Blood pressure difference
* Proportions of patients with BP reached the target (130/80 mmHg)
* Number of anti-hypertensive drugs use to achieve BP target
* Urine albumin/creatinine ratio
* Major Adverse Cardiac Events (MACE)
* Cardio-ankle vascular index (CAVI)
* ankle-brachial index (ABI)

Documentary Proof of Ethical Clearance :

This project has been reviewed and approved by the Comittee on Human Rights Related to Research Involving Human Subjects , based on the declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3-4 (eGFR 15-59 mL/min/1.73m²)
* Microalbuminuria
* Any blood pressure level

Exclusion Criteria:

* Salt - losing conditions
* Hyponatremia (Na < 135 mg/dL) or Hypernatremia (Na > 145 mg/dL)
* Bilateral renal artery stenosis
* Severe comorbid disease or life expectancy <1 year (severe cardiovascular disease, chronic liver disease, severe infection , malignancy)
* Immunosuppressant used

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The declination of glomerular infiltration rate | one year